CLINICAL TRIAL: NCT04759196
Title: Generating Evidence on NonEpileptic, Stereotypical and Intermittent Symptoms (NESIS) in Chronic Subdural Hematomas
Acronym: GENESIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-31-2021-3687
Record Dates: First submitted 2020-10-27; First posted 2021-02-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Subdural Hematoma; Epilepsy; Seizure; Cortical Depression; Cortical Depolarization; Nonepileptic, Stereotypical and Intermittent Symptoms; NESIS
Keywords: Transient neurological symptoms; Levetiracetam; keppra; Lamotrigine; lamictal
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Epilepsy | interventions — Topiramate; Levetiracetam

STUDY DESIGN:
Intervention Model Description: Patients with chronic subdural hematomas, transient neurological symptoms with negative EEG will be divided in two groups based on their NESIS scores (up to 3 (increased risk of epileptic seizures) and 4 or more (increased risk of cortical depression)). Those two groups are going to receive both Levetiracetam or Lamotrigine.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participant will not know the medication they are taking. When accepting to participate, they are going to have the full list of possible side effects, without knowing which one are link to which medication.
  The doctors in charge of administering the questionnaires will be blind. The person in charge of analyzing the results will also be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NESIS - Levetiracetam (Active Comparator): Participant with a score NESIS of 4 or more (increased risk of having cortical depression).
  Levetiracetam is an anti-epileptic drug known to be inefficient in other condition with cortical depression. It will be use as an active comparator.
  Interventions: Drug: Levetiracetam
- NESIS - Topiramate (Experimental): Participant with a score NESIS of 4 or more (increased risk of having cortical depression).
  Topiramate is an anti-epileptic drug known to be efficient in other condition with cortical depression. The investigators want to test his efficacy in chronic subdural hematoma with probable cortical depression.
  Interventions: Drug: Topamax
- Non NESIS - Levetiracetam (Active Comparator): Participant with a score NESIS of 3 or less (increased risk of having epileptic discharges).
  Levetiracetam is an anti-epileptic drug known to be inefficient in other condition with cortical depression. It will be use as an active comparator.
  Levetiracetam should be as efficient as Topiramate in a group a participant with epileptic discharges.
  Interventions: Drug: Levetiracetam
- Non-NESIS - Topiramate (Experimental): Participant with a score NESIS of 3 or less (increased risk of having epileptic discharges).
  Topiramate is an anti-epileptic drug known to be efficient in other condition with cortical depression. The investigators want to test his efficacy in chronic subdural hematoma with probable cortical depression.
  Topiramate should be as efficient as Levetiracetam in a group a participant with epileptic discharges.
  Interventions: Drug: Topamax

INTERVENTIONS:
Drug: Topamax — TPM : 50 mg BID, with increased of 50 mg by week until efficacy, to a maximum of 100 mg BID.
  Other Names: Topiramate; TPM
  Arms: NESIS - Topiramate; Non-NESIS - Topiramate
Drug: Levetiracetam — LEV : 500 mg BID, with increase of 1000 mg die divided in two doses each week until efficacy, to a maximum of 1500 mg BID.
  Other Names: LEV; Keppra
  Arms: NESIS - Levetiracetam; Non NESIS - Levetiracetam

SUMMARY:
Some patients with chronic subdural hematomas and transient neurological symptoms do not respond to standard antiepileptic drugs. The investigators think that some of them could have cortical depression rather than epileptic discharges. After an intensive literature review, the investigators found out that some antiepileptic dugs (Lamotrigine, Topiramate) were found to be efficient to treat cortical depression in other conditions (migraine, subarachnoid hemorrhage). In contrast, some other drugs (Levetiracetam) were not proved to be efficient. Knowing that, the investigators want to compare the efficacy of Topiramate against Levetiracetam in two different groups, the NESIS group (based on a NESIS score of 4 or more - increased risk of cortical depression) versus a non-NESIS group (score of 3 or less - increased risk of epileptic discharges).

DETAILED DESCRIPTION:
Patients presenting with transient neurological symptoms in the context of subdural hemorrhage may present a diagnostic challenge. Many of these patients end up with a probable diagnosis of epilepsy (or acute symptomatic seizures), despite a negative electroencephalogram. The investigators believe that the origin of these transient neurologic symptoms in a significant subpopulation of these patients may in fact be cortical depolarization, rather than epileptiform activity. Very specific characteristics have already been identified that differentiate these patients from those who ultimately have epilepsy. The NESIS entity (nonepileptic, stereotypical, and intermittent symptoms) has been proposed to represent this group of patients. A NESIS score was then designed to help distinguish patients with epileptiform activity (confirmed by EEG) from those likely to have cortical depolarization. In other diseases presenting cortical depolarizations, certain antiepileptic treatments (including Topiramate) have already been recognized as effective. The investigators therefore want to perform a prospective, multicenter, randomized-controlled study (Topiramate group and Levetiracetam group) to determine whether a significant difference in the response to treatment exists between Topiramate and Levetiracetam in the NESIS group compared to the non-NESIS group. In addition, in a few eligible patients, the investigators will implant an electrocorticography electrode to demonstrate the existence of cortical depolarizations.

ELIGIBILITY:
Inclusion Criteria:

* Be aged ≥ 18 years
* Chronic subdural hematoma
* Transient neurological symptoms (Sensory, motor, cerebellar or speech symptoms, lasting 6 hours or less)
* Initial negative EEG

Exclusion Criteria:

* Contraindications to Levetiracetam
* Psychiatric history (major depression, psychosis, risk of suicide)
* History of hypersensitivity to LEV (anaphylaxis, angioedema, skin reaction)
* Contraindications to Topiramate
* History of hypersensitivity to TPM
* Glaucoma
* Past of nephrolithiasis
* Known epilepsy or past seizure before the current subdural hemorrhage
* Actual taking of an antiepileptic drug
* Intracranial pathology not caused by subdural hematoma (intra-parenchymal hemorrhage, neoplasia)
* Pregnancy or planning to
* Inability to carry out the necessary follow-ups for the study
* Refusal of the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in the number of TNS reported at 6 month in participants with a positive Nonepileptic, Stereotyped, Intermittent Symptoms (NESIS) score (4 and more) | Through study completion, an average of 3 years
  The aim of this study is to demonstrate the efficacy of Topiramate in the treatment of patients with transient neurological symptoms in the context of chronic subdural hemorrhage with a positive NESIS score (4 and more), in whom usual epilepsy treatment appears to be less effective. To do this, the effect of Topiramate (shown to be effective in cortical depressions) will be compared with that of Levetiracetam (which has not been shown to be effective in cortical depressions). This is going to be done by a questionnaire that will assess the resolution of symptoms or not, or the percentage of diminution.

SECONDARY OUTCOMES:
Between-group difference in the number of TNS reported at 6 month in all participants (all NESIS scores) | Through study completion, an average of 3 years
  If the investigators manage to demonstrate a significant difference between the response to TPM and LEV in the NESIS group compared to the non-NESIS group with our questionnaire, the evidence concerning the existence of a different process at the origin of the NESIS group will then be more numerous. As demonstrated in studies on rats, cortical spreading depolarization respond well to TPM and not to LEV. Cortical depolarizations will then be the main hypothesis of the reason why some responds better to TPM than LEV in our study.
Incidence of cortical spreading depression on electrocorticography in the first postoperative week of patients with preoperative TNS. | Through study completion, an average of 3 years
  The investigators think that cortical depression rather then epileptic discharges could be involved in some patients with transient neurological symptoms in context of subdural hematomas. Some participant could need decompression surgery for their subdural hematoma. The investigators will offer the insertion of electrocorticography electrods while this surgery. The aim of this intervention will be to prove cortical depression in some subjects by using electrocorticography that will be read by a neurologist specialized in epilepsy.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Iorio-Morin, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cousseau DH, Echevarria Martin G, Gaspari M, Gonorazky SE. [Chronic and subacute subdural haematoma. An epidemiological study in a captive population]. Rev Neurol. 2001 May 1-15;32(9):821-4. Spanish. PMID 11424031
- [Background] Toi H, Kinoshita K, Hirai S, Takai H, Hara K, Matsushita N, Matsubara S, Otani M, Muramatsu K, Matsuda S, Fushimi K, Uno M. Present epidemiology of chronic subdural hematoma in Japan: analysis of 63,358 cases recorded in a national administrative database. J Neurosurg. 2018 Jan;128(1):222-228. doi: 10.3171/2016.9.JNS16623. Epub 2017 Feb 3. PMID 28156246
- [Background] Won SY, Dubinski D, Herrmann E, Cuca C, Strzelczyk A, Seifert V, Konczalla J, Freiman TM. Epileptic Seizures in Patients Following Surgical Treatment of Acute Subdural Hematoma-Incidence, Risk Factors, Patient Outcome, and Development of New Scoring System for Prophylactic Antiepileptic Treatment (GATE-24 score). World Neurosurg. 2017 May;101:416-424. doi: 10.1016/j.wneu.2017.02.024. Epub 2017 Feb 16. PMID 28213197
- [Background] King MA, Newton MR, Jackson GD, Fitt GJ, Mitchell LA, Silvapulle MJ, Berkovic SF. Epileptology of the first-seizure presentation: a clinical, electroencephalographic, and magnetic resonance imaging study of 300 consecutive patients. Lancet. 1998 Sep 26;352(9133):1007-11. doi: 10.1016/S0140-6736(98)03543-0. PMID 9759742
- [Background] Levesque M, Iorio-Morin C, Bocti C, Vezina C, Deacon C. Nonepileptic, Stereotypical, and Intermittent Symptoms (NESIS) in Patients With Subdural Hematoma: Proposal for a New Clinical Entity With Therapeutic and Prognostic Implications. Neurosurgery. 2020 Jul 1;87(1):96-103. doi: 10.1093/neuros/nyz355. PMID 31555809
- [Background] Woitzik J, Hecht N, Pinczolits A, Sandow N, Major S, Winkler MK, Weber-Carstens S, Dohmen C, Graf R, Strong AJ, Dreier JP, Vajkoczy P; COSBID study group. Propagation of cortical spreading depolarization in the human cortex after malignant stroke. Neurology. 2013 Mar 19;80(12):1095-102. doi: 10.1212/WNL.0b013e3182886932. Epub 2013 Feb 27. PMID 23446683
- [Background] Klass A, Sanchez-Porras R, Santos E. Systematic review of the pharmacological agents that have been tested against spreading depolarizations. J Cereb Blood Flow Metab. 2018 Jul;38(7):1149-1179. doi: 10.1177/0271678X18771440. Epub 2018 Apr 20. PMID 29673289
- [Background] Harriott AM, Takizawa T, Chung DY, Chen SP. Spreading depression as a preclinical model of migraine. J Headache Pain. 2019 May 2;20(1):45. doi: 10.1186/s10194-019-1001-4. PMID 31046659
- [Background] Shank RP, Gardocki JF, Streeter AJ, Maryanoff BE. An overview of the preclinical aspects of topiramate: pharmacology, pharmacokinetics, and mechanism of action. Epilepsia. 2000;41(S1):3-9. PMID 10768292
- [Background] Bagnato F, Good J. The Use of Antiepileptics in Migraine Prophylaxis. Headache. 2016 Mar;56(3):603-15. doi: 10.1111/head.12781. Epub 2016 Mar 3. PMID 26935348
- [Background] Ashtari F, Shaygannejad V, Akbari M. A double-blind, randomized trial of low-dose topiramate vs propranolol in migraine prophylaxis. Acta Neurol Scand. 2008 Nov;118(5):301-5. doi: 10.1111/j.1600-0404.2008.01087.x. PMID 18713156
- [Background] Storey JR, Calder CS, Hart DE, Potter DL. Topiramate in migraine prevention: a double-blind, placebo-controlled study. Headache. 2001 Nov-Dec;41(10):968-75. doi: 10.1046/j.1526-4610.2001.01190.x. PMID 11903524
- [Background] Brandes JL, Saper JR, Diamond M, Couch JR, Lewis DW, Schmitt J, Neto W, Schwabe S, Jacobs D; MIGR-002 Study Group. Topiramate for migraine prevention: a randomized controlled trial. JAMA. 2004 Feb 25;291(8):965-73. doi: 10.1001/jama.291.8.965. PMID 14982912
- [Background] Millan-Guerrero RO, Isais-Millan R, Barreto-Vizcaino S, Gutierrez I, Rivera-Castano L, Trujillo-Hernandez B, Baltazar LM. Subcutaneous histamine versus topiramate in migraine prophylaxis: a double-blind study. Eur Neurol. 2008;59(5):237-42. doi: 10.1159/000115637. Epub 2008 Feb 8. PMID 18264012
- [Background] Diener HC, Tfelt-Hansen P, Dahlof C, Lainez MJ, Sandrini G, Wang SJ, Neto W, Vijapurkar U, Doyle A, Jacobs D; MIGR-003 Study Group. Topiramate in migraine prophylaxis--results from a placebo-controlled trial with propranolol as an active control. J Neurol. 2004 Aug;251(8):943-50. doi: 10.1007/s00415-004-0464-6. PMID 15316798
- [Background] Mei D, Capuano A, Vollono C, Evangelista M, Ferraro D, Tonali P, Di Trapani G. Topiramate in migraine prophylaxis: a randomised double-blind versus placebo study. Neurol Sci. 2004 Dec;25(5):245-50. doi: 10.1007/s10072-004-0350-0. PMID 15624081
- [Background] Silberstein SD, Neto W, Schmitt J, Jacobs D; MIGR-001 Study Group. Topiramate in migraine prevention: results of a large controlled trial. Arch Neurol. 2004 Apr;61(4):490-5. doi: 10.1001/archneur.61.4.490. PMID 15096395
- [Background] Gupta P, Singh S, Goyal V, Shukla G, Behari M. Low-dose topiramate versus lamotrigine in migraine prophylaxis (the Lotolamp study). Headache. 2007 Mar;47(3):402-12. doi: 10.1111/j.1526-4610.2006.00599.x. PMID 17371357
- [Background] Beran RG, Spira PJ. Levetiracetam in chronic daily headache: a double-blind, randomised placebo-controlled study. (The Australian KEPPRA Headache Trial [AUS-KHT]). Cephalalgia. 2011 Apr;31(5):530-6. doi: 10.1177/0333102410384886. Epub 2010 Nov 8. PMID 21059626
- [Background] Linde M, Mulleners WM, Chronicle EP, McCrory DC. Antiepileptics other than gabapentin, pregabalin, topiramate, and valproate for the prophylaxis of episodic migraine in adults. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD010608. doi: 10.1002/14651858.CD010608. PMID 23797674
- [Background] Unekawa M, Tomita Y, Toriumi H, Suzuki N. Suppressive effect of chronic peroral topiramate on potassium-induced cortical spreading depression in rats. Cephalalgia. 2012 May;32(7):518-27. doi: 10.1177/0333102412444015. Epub 2012 Apr 20. PMID 22523186
- [Background] Akerman S, Goadsby PJ. Topiramate inhibits cortical spreading depression in rat and cat: impact in migraine aura. Neuroreport. 2005 Aug 22;16(12):1383-7. doi: 10.1097/01.wnr.0000175250.33159.a9. PMID 16056144
- [Background] Ayata C, Jin H, Kudo C, Dalkara T, Moskowitz MA. Suppression of cortical spreading depression in migraine prophylaxis. Ann Neurol. 2006 Apr;59(4):652-61. doi: 10.1002/ana.20778. PMID 16450381
- [Background] Lin CH, Hsu SP, Cheng TC, Huang CW, Chiang YC, Hsiao IH, Lee MH, Shen ML, Wu DC, Zhou N. Effects of anti-epileptic drugs on spreading depolarization-induced epileptiform activity in mouse hippocampal slices. Sci Rep. 2017 Sep 19;7(1):11884. doi: 10.1038/s41598-017-12346-y. PMID 28928441
- [Background] Abou-Khalil BW. Update on Antiepileptic Drugs 2019. Continuum (Minneap Minn). 2019 Apr;25(2):508-536. doi: 10.1212/CON.0000000000000715. PMID 30921021
- [Background] Zhuo C, Jiang R, Li G, Shao M, Chen C, Chen G, Tian H, Li J, Xue R, Jiang D. Efficacy and Tolerability of Second and Third Generation Anti-epileptic Drugs in Refractory Epilepsy: A Network Meta-Analysis. Sci Rep. 2017 May 31;7(1):2535. doi: 10.1038/s41598-017-02525-2. PMID 28566726
- See also: Topiramate. Drug information. — https://www.uptodate.com/contents/topiramate-drug-information?search=topiramate&usage_type=panel&kp_tab=drug_general&source=panel_search_result&selectedTitle=1~148&display_rank=1
- See also: Levetiracetam. Drug information. — https://www.uptodate.com/contents/levetiracetam-drug-information?search=keppra&source=panel_search_result&selectedTitle=1~82&usage_type=panel&kp_tab=drug_general&display_rank=1
- See also: Santé canada, registres des produits pharmaceutiques. (Canadian drugs register) — https://hpr-rps.hres.ca/details.php?drugproductid=636&query=APO-TOPIRAMATE
- See also: Side effects classification — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_8.5x11.pdf

DOCUMENTS (2):
  • Study Protocol (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04759196/Prot_000.pdf
  • Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04759196/ICF_001.pdf